CLINICAL TRIAL: NCT05098002
Title: Mindfulness Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 1946021
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful based stress classes (Experimental): 6 week mindfulness program
  Interventions: Behavioral: Mindfulness program

INTERVENTIONS:
Behavioral: Mindfulness program — 6 week class designed to improve psychological well-being

SUMMARY:
To offer Roswell Park patients and caregivers a variety of options to reduce their stress and improve their psychological well-being amidst the difficulty of cancer

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Cancer survivor or a caregiver of cancer patient/survivor.

Exclusion Criteria:

* Unwilling or unable to complete the assessment in English.
* Are unwilling or unable to follow protocol requirements.
* Have any condition which in the Investigator's opinion deems the subject an unsuitable candidate to participate in this study including (based on criteria from the Mindfulness-based stress reduction (MBSR) authorized curriculum guide):

  1. Drug addiction (or recent recovery)
  2. Bereavement (recent loss)
  3. Mental health inpatient (recently discharged)
  4. Current depression or other major psychiatric diagnoses (including suicidality or suicidal ideation) that would interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Feasibility - Enrollment rates | 6 weeks
  Number of participants enrolled in virtual classes vs in person classes

SECONDARY OUTCOMES:
Acceptability | 6 weeks
  Percentage of participants who choose in person classes vs. virtual classess

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided